CLINICAL TRIAL: NCT05979649
Title: The Effectiveness of an Internet-Based Intervention With Peer Support for the Mental Health of Youths: A Randomized Controlled Trial
Brief Title: An Internet-Based Intervention With Peer Support for the Mental Health of Youths
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wei XIA, PhD (Other)
Responsible Party: Sponsor-Investigator, Wei XIA, PhD, Associate Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: L2023SYSU-HL-010
Record Dates: First submitted 2023-07-29; First posted 2023-08-07 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Mental Health Issue
Keywords: adolescent; internet-based; peer support; post-pandemic era; stressful life event; Coping Behavior

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- experimental group (Experimental): 1. Throughout the intervention period, we will deliver weekly customized feeds to youths at a consistent time, covering stressful events, coping strategies, social support, and emotional intelligence, totaling eight deliveries.
  2. After peer interveners (peer mentors) receive counseling credentials, every fifth participant will be randomly paired with a peer intervener. Over the next eight weeks, they will engage in individualized conversations via online video conferences biweekly.The intervention will last eight weeks, with four conversations in total.
  3. After each personalized conversation, the interveners will collaboratively develop behavioral corrective tasks for the following two weeks from the "To Do List," including at least one task from each category: social support, coping strategies, and emotional intelligence. During the next conversation, the interveners will inquire about the participants' completion status and personal experiences.
  Interventions: Behavioral: behavioral corrective tasks; Other: Counselling on psychological knowledge
- control group (Placebo Comparator): Throughout the eight weeks of intervention, articles without professional psychological knowledge will be delivered to the control group participants once a week at a consistent time, totaling eight deliveries in total.
  Interventions: Other: placebo-controlled study
- Peer intervener group (Other): Peer interveners will participate in a one-day course conducted by several instructors with backgrounds in psychology and medicine. They will be required to pass a "standardized patient test" after the course to obtain the qualification for intervention.
  Interventions: Other: Peer Interventionist Training

INTERVENTIONS:
Behavioral: behavioral corrective tasks — After each personalized conversation, the interveners will, based on a clear understanding of the participants' completion status and personal experiences with the previous "behavioral corrective tasks," assist in formulating future "behavioral corrective tasks" for the next two weeks. These tasks will be selected from our designated "To Do List," requiring at least one task from each category: social support, coping strategies, and emotional intelligence.
  Arms: experimental group
Other: Counselling on psychological knowledge — Counselling on psychological knowledge includes weekly personalized feeds, as well as the methods and techniques for coping with challenges provided by the interveners.during personalized conversations with the participants.
  Arms: experimental group
Other: placebo-controlled study — "feel-good" articles without professional psychological knowledge will be sent to the control group participants weekly.
  Arms: control group
Other: Peer Interventionist Training — The training is a one-day course, encompassing a broad range of topics, including but not limited to counseling techniques and specialized medical psychology knowledge.
  Arms: Peer intervener group

SUMMARY:
The aim of this randomized control trial study is to develop an online intervention project that specifically targets and addresses mental health issues among youths in the post-pandemic era, while also assessing its effectiveness. Additionally, this intervention project has the potential to effectively address other post-traumatic conditions experienced by youths. Furthermore, our research group will investigate the specific impacts of long-term interventions on various aspects including changes in mental health status, psychological resilience, coping strategies, perceived social support, and emotional intelligence among the participants.

DETAILED DESCRIPTION:
Over the past decade, mental health issues have become increasingly prevalent among young people. Approximately 14% of adolescents aged 10-19 years globally suffer from conditions like depression and anxiety. This is concerning because adolescence is a critical period for development, and these mental health problems can have long-term consequences on various aspects of their lives, including relationships, education, and work.

The mental health of young people (15-24) is a significant global concern, affecting one in five individuals within this age group and representing the largest burden of illness. Moreover, the impact of mental health problems during adolescence can extend into adulthood, affecting physical and mental well-being and limiting opportunities for a fulfilling life.

According to the World Health Organization (WHO), mental health and psychosocial well-being are essential for youth's human potential and rights. However, the COVID-19 pandemic has exacerbated mental health problems among adolescents, leading to disruptions in critical mental health services in many countries. Studies have shown that the pandemic has resulted in increased depression, anxiety, stress, and sleep disorders among young people. Additionally, the previously mentioned conditions faced by adolescents have worsened to the point of mental disorders and suicide attempts.

The impact of the pandemic on youths' mental health has drawn global attention and highlights the urgency of intervening in their mental well-being. Stressors among young people primarily come from academics, employment, relationships, appearance, finances, etc. The lack of effective coping strategies and emotional regulation further exacerbate physical health symptoms and negative consequences. Unfortunately, a significant number of young people experiencing mental health problems do not seek professional help, primarily due to denial, embarrassment, lack of time, and stigma. They often turn to informal resources such as family, friends, books, or counseling websites, with uncertain effectiveness. Long waiting lists for psychological services add to the dilemma. Therefore, it is crucial to help youths overcome these barriers when providing support services.

Currently, access to cost-effective and accessible mental health services remains challenging for young people. In addition to counseling and psychiatric services, peer support has emerged as a novel resource for young people seeking help. Peer support involves social and emotional support from individuals with similar experiences. Research suggests that peer support is an accessible, affordable, and easily implemented mental health resource. Involving peer supporters in mental health services can promote recovery and has positive effects on depressive symptoms, anxiety, psychological distress, self-esteem, self-efficacy, and self-management. However, there is a lack of research on the development and implementation of peer-support based interventions for adolescents with psychological problems. This study aims to address this gap.

Given the concerns surrounding psychological problems among young people, this study aims to design a pragmatic and comprehensive peer support-based intervention. The intervention will be based on the Youth Stressful Life Event Response Model, which explains how adolescents respond to stress and how factors like emotional intelligence, social support, and coping strategies impact their mental health. This online, single-blind, randomized controlled trial will include both an intervention group and a control group. The control group will receive motivational articles unrelated to the main monitoring indicators. Participants will be assessed at baseline, post-intervention, and during follow-up. Through the implementation of a peer support program, this study aims to investigate the specific effects of long-term intervention on changes in mental health status, psychological resilience, perceived social support, and emotional intelligence.

ELIGIBILITY:
Experimental group and control group:

Inclusion Criteria:

* Aged 14-25
* Individuals who have experienced a stressful life event of moderate or greater magnitude within the past six months (with a moderate impact on one or more of the Stressful Events Scale screenings).
* Individuals who can provide informed consent and willingly cooperate with this study

Exclusion Criteria:

* Individuals currently undergoing clinical psychotherapy or participating in other interventional studies.
* Individuals diagnosed with psychological or mental disorders.

Peer intervener group：

Inclusion Criteria:

* Aged 18-25
* Individuals with a Bachelor's degree in progress or higher, and a professional background in sociology, psychology, education, or medicine.
* Individuals who can provide informed consent and willingly cooperate with this study.

Exclusion Criteria:

* Individuals currently undergoing clinical psychotherapy or participating in other interventional studies.
* Individuals diagnosed with psychological or mental disorders.

Ages: 14 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
The ability to cope with stressful situations | Baseline,2 months，4 months
  The change of the scores of various dimensions in the Stressful Situation Coping Scale - Chinese short(CISS-SFC) among youths during the intervention period and follow-up period.This scale is divided into four dimensions: task-oriented coping, emotion-oriented coping, distraction coping, and social diversion coping.Each item consists of four statements (scoredfrom 0 to 3) describing depressive symptoms, with higher scores indicating greater severity. Scores on eachitem are summed to yield a total score on the measure from 0 to 63.
The level of emotional intelligence | Baseline,2 months，4 months
  The change of the Wong and Law Emotional Intelligence Scale(WLEIS) scores of youths during the intervention and follow-up periods.This scale includes four sub-scales: appraisal and expression of emotion in oneself, appraisal and recognition of emotion in others, regulation of emotion in oneself, and use of emotion to facilitate performance.The scale score ranges from 16 to 112.The higher the score, the better the emotional intelligence of youths.
The mental health level of the youths | Baseline,2 months，4 months
  The change of the Brief Symptom Inventory-53(BSI-53) scores of youths during the intervention and follow-up periods.The minimum score on the scale is 0.The sum of all items' scores reaching 63 and above was considered "BSI-positive" .The lower the score, the milder the psychological problem symptoms of youths.
The participants' somatization symptoms, anxiety, and depression status | Baseline,2 months，4 months
  The change of the Brief Symptom Inventory-18(BSI-18) scores of youths during the intervention and follow-up periods.The scale has a minimum score of 0 and a maximum score of 72. The higher the score, the worse the psychological well-being of adolescents.
The perceived level of social support system for oneself | Baseline,2 months，4 months
  The change of the Perceived Social Support Scale(PSSS) scores during the intervention and follow-up periods.The scale score ranges from 7 to 84, and the higher the score, the greater the perceived level of social support by the participants.
Subjects' mental toughness Connor-Davidson resilience scale | Baseline,2 months，4 months
  The change of the Connor-Davidson resilience scale scores during the intervention and follow-up periods.The scale has a minimum score of 0 and a maximum score of 100. The higher the score, the better the psychological resilience of the participants.

SECONDARY OUTCOMES:
The extent of negative impact caused by stressful life events. | Baseline,2 months，4 months
  The change of the Adolescent Self-Rating Life Events Check-List scale(ASLEC) scores of youths during the intervention period and follow-up period.The scores on the scale range from 0 (with the lowest score being 3 for participants meeting the inclusion criteria of this study) to 135. A higher score indicates a greater impact of stressful life events on the participants.
The level of social support received. Social Support Rating Scale | Baseline,2 months，4 months
  The change of the Social Support Rating Scale(SSRS) scores during the intervention and follow-up periods.This scale includes objective support, subjective support, and utilization of support.The sum of all scores from the three subscales to obtain aggregate scores for the SSRS. A higher score indicates a higher level of social support.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Xia, PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- XIAW, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
The non-identified IPD will be shared after the outcomes have been published.
Supporting Information: SAP
Time Frame: After the publication of the study
Access Criteria: Researchers should contact the PI for approval of the study protocol.